CLINICAL TRIAL: NCT07242976
Title: Evaluation of Balance Using the Biodex Balance System Among Different Subcategories of Low Back Pain
Acronym: Biodex
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Delta University for Science and Technology (Other)
Responsible Party: Principal Investigator, Muhammed El-sayed Muhammed Abu l Ftouh, Demonstrator at orthopedic department faculty of physical therapy delta university, Delta University for Science and Technology
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: BIODEX BALANCE SYSTEM
Record Dates: First submitted 2025-11-14; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain; Spondylolisthesis; Spondylosis Lumbar; Balance Assessment
Keywords: biodex; balance; subcategories of low back pain
MeSH Terms: conditions — Low Back Pain; Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index (APSI), and overall stability index (OSI). Each index is further measured in four outcomes: Double leg eyes open (DLEO), Double leg eyes closed (DLEC), Single leg eye open (SLEO) for both legs and Single leg eye closed (SLEC) for both legs. Additionally Biodex Balance Systen (BBS) will assess limit of stability in one outcome: Double leg eyes open (DLEO).
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group (GI)= will include 20 healthy normal subjects. (Active Comparator): Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index (APSI), and overall stability index (OSI). Each index is further measured in four outcomes: Double leg eyes open (DLEO), Double leg eyes closed (DLEC), Single leg eye open (SLEO) for both legs and Single leg eye closed (SLEC) for both legs. Additionally Biodex Balance Systen (BBS) will assess limit of stability in one outcome: Double leg eyes open (DLEO).
  Interventions: Diagnostic Test: Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index
- Group (GII) will include 20 patients with lumbar spondylosis. (Active Comparator): Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index (APSI), and overall stability index (OSI). Each index is further measured in four outcomes: Double leg eyes open (DLEO), Double leg eyes closed (DLEC), Single leg eye open (SLEO) for both legs and Single leg eye closed (SLEC) for both legs. Additionally Biodex Balance Systen (BBS) will assess limit of stability in one outcome: Double leg eyes open (DLEO).
  Interventions: Diagnostic Test: Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index
- Group (GIII) will include 20 patients with lumbar spondylolisthesis. (Active Comparator): Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index (APSI), and overall stability index (OSI). Each index is further measured in four outcomes: Double leg eyes open (DLEO), Double leg eyes closed (DLEC), Single leg eye open (SLEO) for both legs and Single leg eye closed (SLEC) for both legs. Additionally Biodex Balance Systen (BBS) will assess limit of stability in one outcome: Double leg eyes open (DLEO).
  Interventions: Diagnostic Test: Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index
- Group (GIV) will include 20 patients with lumbar disc prolapse. (Active Comparator): Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index (APSI), and overall stability index (OSI). Each index is further measured in four outcomes: Double leg eyes open (DLEO), Double leg eyes closed (DLEC), Single leg eye open (SLEO) for both legs and Single leg eye closed (SLEC) for both legs. Additionally Biodex Balance Systen (BBS) will assess limit of stability in one outcome: Double leg eyes open (DLEO).
  Interventions: Diagnostic Test: Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index

INTERVENTIONS:
Diagnostic Test: Assessment of balance will be measured by The Biodex Balance System (BBS) which computes Postural Stability key indices: the medial-lateral stability index (MLSI), anterior-posterior stability index — Low back pain (LBP) is a leading cause of disability worldwide and is often associated with postural and balance impairments. However, limited evidence exists on how these deficits differ among specific types of LBP such as lumbar spondylosis, spondylolisthesis, and disc prolapse. Understanding these variations is crucial for accurate assessment and targeted rehabilitation. Evaluating balance using the Biodex Balance System can help identify the extent of impairment and guide physiotherapists in developing individualized rehabilitation programs that enhance postural control, stability, and functional performance, ultimately improving quality of life and reducing fall risk among LBP patients.
  Other Names: Arabic Numerical Rating Scale; Arabic version of Oswestry disability index (Ar-ODI)

SUMMARY:
this study aims to evaluate balance using the biodex balance system among patients with spondylosis, spondylolisthesis, and lumber disc prolapse.

DETAILED DESCRIPTION:
Low back pain is one of the most common causes of disability globally . While postural balance impairments have been widely documented in individuals with low back pain, there is limited understanding of how these impairments vary across specific subcategories of specific low back pain. Low back pain is generally categorized into non specific and specific types.

Non-specific LBP approximately accounts for 85-90% of all low back pain cases (Hartvigsen et al., 2018). In contrast, specific low back pain arises from a recognizable pathology such as structural abnormalities. The most common causes of specific low back pain are lumbar spondylosis, spondylolisthesis, and lumbar disc prolapse. Lumbar spondylosis has a prevalence of 74% in individuals over 60 years confirmed with radiographic findings. Spondylolisthesis affects approximately 6-11.5% of adults , lumbar disc prolapse accounts for 2-5% of all low back pain cases.

Balance deficiency among patients with spondylosis, spondylolisthesis and lumber disc prolapse was reported in literature by different objective assessment tools. Individuals with low back pain exhibit measurable deficits in balance and postural stability compared to healthy controls . Also, the chronicity of low back pain affects both static and dynamic balance.

Assessment and detection of balance deficiency among patients with spondylosis, spondylolisthesis and lumber disc prolapse will allow physical therapists to design individualized rehabilitation programs. Improve understanding of interventions focusing on core stabilization, proprioceptive retraining and dynamic balance. This may improve postural control, enhance gait performance, reduce fall risk and support better functional outcomes in daily activities.

Thus, there was a need to study the difference in balance using the biodex balance system among patients with spondylosis, spondylolisthesis and lumber disc prolapse. The current study may provide a more conclusive insight in evaluation and treatment of patients with low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic low back pain (≥3 months duration) (Ge et al., 2021). Referred from orthopedic surgeons with confirmed diagnosis of lumbar spondylosis, spondylolisthesis or lumber disc prolapse affecting L4-L5 or L5 S1( Hlaing et al., 2020) depending on imaging findings (MRI, CT or X-ray scan within the last 6 months):

  * Lumbar spondylosis; defined as degenerative disc disease, osteophyte formation with or without facet joint arthropathy (Natarajan et al., 2021; Christe et al., 2020).
  * Lumbar spondylolisthesis; defined as anterolisthesis of one vertebral body over another, graded via the Meyerding scale (grade 1 or 2) (Giordan et al., 2023; Chuang et al., 2018).
  * Lumbar disc prolapse; defined as protrusion, herniation of intervertebral disc (Kang et al., 2016; Hahne et al., 2019).

    * Age of patients ranges from 35 to 55 years (Albeshri, et.al., 2017)
    * Both genders will be included in the study
    * Pain intensity: ≥ 4/10 on a numerical pain rating scale (Thong et al., 2011).
    * BMI ranged from (18.5-29.9 kg/m²) (Karimi et al., 2008; Soliman et al., 2017).
    * Healthy subjects are healthy volunteers and without any Musculoskeletal disorders (Karimi et al., 2008).

Exclusion Criteria:

* The following patients will be excluded from the study patients with:

  * Prior lumbar spine surgery or neurological disorders (e.g., parkinson's, stroke) that may influence balance (soliman et al., 2017).
  * Fractures of the spine, pelvis or lower extremities, (Karimi et al., 2008).
  * Leg length discrepancy(Karimi et al., 2008).
  * Systemic disease such as arthritis, tuberculosis, liver or kidney failure. (Karimi et al., 2008).
  * Patients with chronic non-specific low back pain.
  * Patients exhibiting red flag symptoms such as urinary or fecal incontinence, saddle anesthesia, progressive motor deficits (e.g., foot drop), or other signs of serious neurological compromis (Ruhe et al., 2011).
  * Participants experiencing low back pain with pain radiating distaly below the level of knee (Hlaing et al., 2020).

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Postural stability ( Overall Stability Index) | All postural assessments will be performed for 20 seconds
  Postural stability will be assessed using the Biodex Balance System through the Overall Stability Index (OSI).The OSI reflects the degree of platform sway, with lower values indicating better balance control. Measurements will be taken under six standardized conditions to evaluate both static and dynamic balance performance. These conditions include:
  Double-Leg, Eyes Open (DLEO)
  Double-Leg, Eyes Closed (DLEC)
  Single-Leg, Eyes Open (SLEO) - Dominant Leg
  Single-Leg, Eyes Closed (SLEC) - Dominant Leg
  Single-Leg, Eyes Open (SLEO) - Non-Dominant Leg
  Single-Leg, Eyes Closed (SLEC) - Non-Dominant Leg
Postural Stability: Medial-Lateral Stability Index (MLSI) | All postural assessments will be performed for 20 seconds
  The Medial-Lateral Stability Index (MLSI) will be obtained from the Biodex Balance System to assess side-to-side postural control. Higher MLSI values indicate greater medial-lateral sway, while lower values reflect better stability in the frontal plane. the measurement will be in six conditions:
  Double leg eyes open (DLEO), Double leg eyes closed (DLEC), Single leg eye open (SLEO) Dominant leg, Single leg eye closed (SLEC) Dominant leg, Single leg eye open (SLEO) Non-Dominant leg and Single leg eye closed (SLEC) Non-Dominant leg
postural stability: Anterior-Posterior Stability Index (APSI) | All postural assessments will be performed for 20 seconds
  The Anterior-Posterior Stability Index (APSI) will be measured using the Biodex Balance System to evaluate forward-backward postural control. Lower APSI values indicate improved stability in the sagittal plane, whereas higher values reflect increased anterior-posterior sway.
  the measurement will be in six conditions: Double leg eyes open (DLEO), Double leg eyes closed (DLEC), Single leg eye open (SLEO) Dominant leg, Single leg eye closed (SLEC) Dominant leg, Single leg eye open (SLEO) Non-Dominant leg and Single leg eye closed (SLEC) Non-Dominant leg
Limits of Stability | All postural assessments will be performed for 20 seconds
  Limits of Stability will be assessed using the Biodex Balance System to evaluate the participant's ability to intentionally shift their center of gravity toward predefined targets without losing balance. The test measures directional control, reaction time, movement speed, and endpoint accuracy, with higher scores reflecting better dynamic balance and voluntary postural control. the measurement condition will be in Double leg eyes open (DLEO)

SECONDARY OUTCOMES:
Arabic version of Numerical pain rating scale (Ar-NPRS) | Periprocedural
  The Numerical Rating Scale is used to quantify the intensity of a subjective symptom-most commonly pain-on a 0 to 10 scale. A score of 0 represents no pain or no symptom, while a score of 10 indicates the worst imaginable pain or maximum symptom severity. Higher scores reflect a worse outcome, indicating greater intensity.
Arabic version of Oswestry disability index (Ar-ODI) | Periprocedural
  The arabic Oswestry Disability Index is a questionnaire used to assess disability related to low back pain. Scores range from 0 to 100, where 0 indicates no disability and 100 indicates maximum disability. Higher scores represent a worse outcome, reflecting greater functional limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Enas F Yousef, Professor of Physical Therapy, Principal Investigator — Physical Therapy for Musculoskeletal Disorders and Its Surgery, Faculty of Physical Therapy, Cairo University; MOAAZ R RIYAD, Lecturer, Study Director — Lecturer of Department of Physical Therapy for Musculoskeletal Disorders and Its Surgery
Locations (1):
- Faculty of Physical Therapy Delta University, Gamasa, Egypt

IPD SHARING:
Plan to Share IPD: No